CLINICAL TRIAL: NCT00620906
Title: Motion Capture Analysis of Sacroiliac Joint Motion After Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Principal Investigator, Dennis Enix, DC, MBA, Assistant Professor, Logan College of Chiropractic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD0524070094
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Sacroiliac Joint Pain
Keywords: manipulation; manual therapy; Sacroiliac joint; effects on manipulation on sacroiliac joint

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): Manipulation
  Interventions: Procedure: Manipulation

INTERVENTIONS:
Procedure: Manipulation — HVLA manipulation to Sacroiliac Joint

SUMMARY:
The purpose of this study is to examine the effects of manipulation on sacroiliac joint motion using a Polhemus motion capture system.

DETAILED DESCRIPTION:
The Sacroiliac (SI) joint is a diarthrodial joint with the contradictory biomechanical function of transmitting compressive loads from the lumbar spine to the lower extremity while maintaining a nutating motion in the pelvis.

Recent studies identify the Sacroiliac (SI) joints as a significant source of pain in patients with chronic low back pain, contributing up to 27%. Recent studies have demonstrated that historical and physical examination findings and radiological imaging alone are insufficient to diagnose SI joint pain.

The purpose of this study is to examine the effects of manipulation on sacroiliac joint motion using a Polhemus motion capture system. The Absolute angular deviation of sacroiliac joint motion will be assessed during the normal gait cycle with the Polhemus Liberty motion capture system. Six sensors will be attached to specific anatomical landmarks of the pelvis which recorded motion characteristics while walking on a treadmill at 5 mph. The subjects then receive a HVLA manipulation to the SI joint and were retested at the same treadmill speed.

The Motion capture system tracks objects at a speed of 240 updates per second on all sensors simultaneously. The latency of data sampling is less than 4ms; 240 x 60 sec x 8 Sensors totaling 115,200 data points per minute. The system generates and tracks electromagnetic fields (EMF), computes position and orientation of sensors in an X, Y, and Z coordinate system while interfacing with a computer. The EMF source contains electromagnetic coils that emit a magnetic field. The source is the system's reference frame for sensor measurements. The sensor contains electromagnetic coils (accelerometers) that detect the position and orientation of the magnetic fields emitted by the EMF source.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 20 and 40
* Ability to maintain normal balance
* Willingness to undergo HVLA manipulation to the SI Joints
* Normal blood pressure

Exclusion Criteria:

* Any visual or vestibular condition or systemic illness that would affect balance
* Any recent surgery, unstable joints of the lower extremity, recent hip and knee joint replacements or fitted hip or knee pins, bolts and/or plates
* Currently have any infection, acute inflammation, recent wounds, injury, tumors or other malignancy
* Currently taking any medications; prescription or herbal muscle stimulants, relaxants, etc.
* A history of acute disc herniation, discopathy or spondylolysis
* A history of acute thrombosis, serious cardiovascular disease, diabetes, have irregular heartbeats(arrhythmia) or wear a pacemaker
* Any implanted device or prosthesis type of device
* Any Spinal manipulation within 48 hours
* Ages under 20 and over 40
* Estimated BMI greater than 30

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Sacroiliac joint motion was assessed with the Polhemus Liberty motion capture system. | Pre and Post therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States